CLINICAL TRIAL: NCT00003064
Title: Phase I-II Study of Tandem Cycles of High Dose Chemotherapy Followed by Autologous Hematopoietic Stem Cell Support in Women With Persistent, Refractory or Recurrent Advanced (Stage III or IV), Epithelial Ovarian Cancer
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Persistent Epithelial Ovarian Cancer, Fallopian Tube, or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065734; CPMC-IRB-7866; NCI-G97-1327; NCT00034320 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Carboplatin; etoposide phosphate; Paclitaxel; Thiotepa; Topotecan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide phosphate
Drug: paclitaxel
Drug: thiotepa
Drug: topotecan hydrochloride
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy and autologous peripheral stem cell transplantation in treating patients with recurrent or persistent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of topotecan with a fixed dose of etoposide phosphate as a component of a multicourse high dose chemotherapy regimen supported by peripheral blood stem cell transplantation in patients with persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.
* Evaluate the response, time to progression, disease free survival, and overall survival in this patient population.

OUTLINE: This is a dose escalation study of topotecan.

All patients receive induction therapy consisting of 1 to 2 courses of mobilization therapy. Subcutaneous filgrastim (G-CSF) is given beginning 24 hours after induction dose. Following induction therapy, peripheral blood stem cells (PBSC) are harvested. After patients receive high dose paclitaxel and carboplatin chemotherapy, a portion of the PBSC are reinfused. When patients recover from the paclitaxel/carboplatin chemotherapy the administration of topotecan and etoposide phosphate begins. Topotecan is administered, as a 72 hour continuous infusion, according to a dose escalation schedule with a fixed dose of etoposide phosphate. A second portion of PBSC are reinfused after topotecan/etoposide phosphate chemotherapy. A course of thiotepa is given along with the final portion of PBSC after treatment with topotecan and etoposide phosphate.

Dose escalation of topotecan continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more patients experience dose limiting toxicity.

Patients are followed every 3 months for 1 year and every 4 months thereafter to determine progression free and overall survival.

PROJECTED ACCRUAL: Approximately 25-30 patients will be accrued for the phase I portion of this study, and 25 more patients will be accrued for the phase II portion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer following at least 3 courses of initial standard platinum based chemotherapy OR have radiologic evidence of recurrence with a CA125 greater than 100
* Initial stage IV disease having a complete response following platinum based therapy allowed
* No brain metastases
* Not eligible for other high priority national or institutional study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Greater than 2 months

Hematopoietic:

* WBC greater than 3000/mm3
* Absolute neutrophil count greater than 1500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT or SGPT less than 1.5 times normal
* PT/PTT within normal limits

Renal:

* BUN less than 1.5 times normal
* Creatinine less than 1.5 times normal
* Creatinine clearance greater than 55 mL/min

Cardiovascular:

* LVEF at least 45%

Other:

* Not pregnant or nursing
* HIV negative
* No prior malignancy other than curatively treated carcinoma in situ of the cervix, nonmelanoma skin cancer, or breast cancer if the risk of recurrence is sufficiently low
* No serious illness that would prevent treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent acetaminophen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Tiersten, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States